CLINICAL TRIAL: NCT01137604
Title: An Open-Label, Three-Cohort, Phase 2 Study of E7080 (Lenvatinib) in Subjects With Recurrent Malignant Glioma
Brief Title: A Study in Subjects With Recurrent Malignant Glioma
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: E7080-G000-203
Record Dates: First submitted 2010-06-02; First posted 2010-06-04 (Estimated); Results first posted 2016-05-23 (Estimated); Last update posted 2022-09-29 (Actual); Status verified 2016-05

CONDITIONS: Glioma
MeSH Terms: conditions — Glioma | interventions — lenvatinib; Bevacizumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): Cohort 1 assessed participants with recurrent Grade 4 malignant glioma (ie, glioblastoma [GBM]) who were bevacizumab-naive. Participants were planned to be accrued in Cohort 1 and randomized in a 1:1 ratio to receive lenvatinib (experimental) or bevacizumab (active comparator).
  Cohort 1 - Bevacizumab
  Cohort 1 - Lenvatinib
  Interventions: Drug: Lenvatinib; Drug: Bevacizumab
- Cohort 2 (Experimental): Cohort 2 assessed participants with recurrent Grade 3 malignant glioma who were bevacizumab-naive. Participants in Cohort 2 were planned to be treated with lenvatinib.
  Interventions: Drug: Lenvatinib
- Cohort 3 (Experimental): Cohort 3 assessed participants with recurrent GBM who had disease progression following prior bevacizumab treatment. Participants in Cohort 3 were planned to be treated with lenvatinib.
  Interventions: Drug: Lenvatinib

INTERVENTIONS:
Drug: Lenvatinib — 24 mg lenvatinib capsules orally, once daily continuously in 28-day cycles until disease progression, development of unacceptable toxicity or withdrawal of consent.
  Other Names: E7080
Drug: Bevacizumab — Bevacizumab 10 mg/kg administered intravenously every 2 weeks in 28-day cycles until disease progression, development of unacceptable toxicity or withdrawal of consent.
  Arms: Cohort 1

SUMMARY:
An open-label phase 2, multicenter study in participants with recurrent malignant glioma.

ELIGIBILITY:
Inclusion Criteria

1. Histologically confirmed diagnosis of Grade 3 or 4 malignant glioma.
2. All subjects who have a first or second recurrence following primary management with surgical resection or biopsy, radiotherapy and up to 2 prior systemic treatments with addition of:

   * No prior bevacizumab treatment is allowed for Cohort 1 and Cohort 2.
   * Subjects must have disease progression following prior bevacizumab treatment for Cohort 3.
   * For all cohorts, no prior anti-vascular endothelial growth factor (VEGF/VEGFR) therapy except for bevacizumab as specified above.
3. Karnofsky score of 70% or greater.
4. Adequately controlled blood pressure (BP) with or without antihypertensive medications, defined as BP less than 150/90 mmHg at screening and no change in antihypertensive medications within 1 week prior to the Screening Visit.
5. Adequate renal function, adequate bone marrow function, adequate blood coagulation function and adequate liver function, as defined in protocol.
6. No evidence of hemorrhage on the baseline magnetic resonance imaging (MRI) scan other than in those subjects who are stable grade 1.

Exclusion criteria:

1. Females who are pregnant or breastfeeding.
2. Subjects who received enzyme-inducing anti-epileptic agents within 14 days before the first dose of study drug (eg, carbamazepine, phenytoin, phenobarbital, primidone, or oxcarbazepine).
3. Active infection requiring intravenous antibiotics.
4. Therapeutic anti-coagulation with warfarin, aspirin, nonsteroidal anti-inflammatory drugs or clopidogrel (low molecular weight heparin is acceptable).
5. Subjects with 24-hour urine protein greater than or equal to 1 gm.
6. Prior surgical resection within 4 weeks, or prior stereotactic biopsy within 2 weeks, of Screening Visit.
7. Prior radiotherapy within 12 weeks unless there is a new area of enhancement consistent with recurrent tumor outside of the radiation field, or there is biopsy-proven unequivocal viable tumor on histopathologic sampling.
8. Prior chemotherapy (6 weeks for nitrosoureas), or any investigational agent within 4 weeks unless the subject has recovered from all anticipated toxicities associated with that therapy; prior bevacizumab therapy (Cohorts 1 and 2); for Cohort 3, prior bevacizumab therapy within 3 weeks.
9. Significant cardiovascular impairment: history of congestive heart failure greater than New York Heart Association (NYHA) Class II ; unstable angina; myocardial infarction or stroke within 6 months of the first dose of study drug; or cardiac arrhythmia requiring medical treatment.
10. Prolongation of QTc interval to greater than 480 msec.
11. Active hemoptysis (bright red blood of at least 1/2 teaspoon) within 3 weeks prior to the first dose of study drug.

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2010-11-09 (Actual); Primary Completion 2013-03-19 (Actual); Study Completion 2014-10-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eisai Medical Services, Study Director — Eisai Inc.
Locations (5):
- United States (3):
  - Tampa, Florida
  - Boston, Massachusetts
  - Durham, North Carolina
- Canada (2):
  - Calgary
  - Toronto

RESULTS

PARTICIPANT FLOW:
Recruitment Details: A total of 173 participants were screened and of those, 152 participants were deemed eligible, and 151 received study treatment.
Pre-assignment Details: The protocol definition of study completion was that the participant had disease progression. Protocol defined reasons for not completing were adverse event, participant choice, lost to follow-up, administrative/other (including withdrawal of consent, pregnancy, study terminated by sponsor or other). Death was not a protocol defined reason for non-completion. Participants were followed for survival until death, except where they withdrew consent, or the Sponsor stopped the survival follow-up.
Groups:
- Cohort 1 - Bevacizumab: Participants with recurrent Grade 4 malignant glioma (ie, glioblastoma [GBM]) who were bevacizumab-naive; received bevacizumab 10 mg/kg administered intravenously every 2 weeks in 28-day cycles
- Cohort 1 - Lenvatinib: Participants with recurrent Grade 4 malignant glioma (ie, glioblastoma [GBM]) who were bevacizumab-naive; received lenvatinib capsules 24 mg taken orally, once daily continuously in 28-day cycles
- Cohort 2 - Lenvatinib: Participants with recurrent Grade 3 malignant glioma who were bevacizumab-naive; received lenvatinib capsules 24 mg taken orally, once daily continuously in 28-day cycles
- Cohort 3 - Lenvatinib: Participants with recurrent GBM who had disease progression following prior bevacizumab treatment; received lenvatinib capsules 24 mg taken orally, once daily continuously in 28-day cycles
Period: Overall Study
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
Started | 38 (39 participants were randomized but 1 participant died prior to receiving treatment.) | 42 | 39 | 32
Treatment Discontinued Due to Disease Progression | 34 | 32 | 26 | 21
Completed | 34 | 32 | 26 | 21
Not Completed | 4 | 10 | 13 | 11
Not completed — Adverse Event | 3 | 6 | 9 | 9
Not completed — Participant Choice | 0 | 2 | 2 | 0
Not completed — Withdrawal of consent | 0 | 0 | 0 | 2
Not completed — Clinical progression/deterioration | 1 | 2 | 2 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib | Total
Number analyzed (Participants) | 38 | 42 | 39 | 32 | 151
Age, Continuous [Mean (Standard Deviation); unit: Years] | 55.1 (10.61) | 55.5 (11.96) | 49.2 (11.35) | 53.0 (11.15) | 52.6 (11.74)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 13 | 10 | 14 | 50
  Male | 25 | 29 | 29 | 18 | 101
World Health Organization Grading for Gliomas [Number; unit: Participants]
  Grade 3 | 0 | 0 | 39 | 0 | 39
  Grade 4 | 38 | 42 | 0 | 32 | 112

OUTCOME MEASURES:

1. Secondary Outcome: Objective Response Rate (ORR)
Description: ORR was the percentage of participants with best overall response (BOR) of complete response (CR) and partial response (PR) based on RANO criteria and investigator's assessment. CR was defined as the disappearance of all enhancing disease (measurable and non-measurable) sustained for at least 4 weeks, no new lesions, and stable or improved non-enhancing (T2/FLAIR) lesions. PR was defined as greater than or equal to 50% decrease, compared to baseline, in the sum of products of perpendicular diameters of all measureable enhancing lesions sustained for at least 4 weeks. No progression of non-measurable disease, no new lesions, stable or improved non-enhancing (T2/FLAIR) lesions on same or lower dose of corticosteroids compared to baseline. For both CR and PR, in the absence of a confirming scan 4 weeks later, this scan was considered only stable disease. Only participants with measureable disease at baseline were included in evaluation of ORR.
Time Frame: From date of randomization (Cohort 1) or first day of treatment (Cohorts 2 and 3) until disease progression, development of unacceptable toxicity, withdrawal of consent or up to data cutoff date of 19 March 2013 (i.e., 2.4 years)
Population: Full Analysis Set included all participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
Number analyzed (Participants) | 38 | 42 | 39 | 32
Percentage of participants | 15.8 [6.0 to 31.3] | 21.4 [10.3 to 36.8] | 7.7 [1.6 to 20.9] | 0.0 [0.0 to 10.9]

2. Secondary Outcome: Progression Free Survival
Description: PFS was measured as the time from randomization (Cohort 1) or the first day of treatment (Cohorts 2 and 3) until the date of first documentation of disease progression or date of death, if death occurred prior to disease progression, based on investigator's assessment.
Time Frame: From date of randomization (Cohort 1) or first day of treatment (Cohorts 2 and 3) until disease progression, development of unacceptable toxicity, withdrawal of consent or up to data cutoff date of 19 March 2013 (ie, 2.4 years)
Population: Full Analysis Set - all participants who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
Number analyzed (Participants) | 38 | 42 | 39 | 32
Months | 2.8 [1.9 to 3.6] | 2.4 [1.8 to 3.6] | 2.8 [1.9 to 3.7] | 1.8 [1.0 to 2.5]

3. Secondary Outcome: Overall Survival (OS)
Description: OS was measured as the time from the randomization date (Cohort 1) or the first day of treatment (Cohort 2 and 3) to the date of death from any cause.
Time Frame: From date of randomization (Cohort 1) or first day of treatment (Cohorts 2 and 3) until death due to any cause or up to data cutoff date of 19 March 2013 (ie, 2.4 years)
Population: Full Analysis Set - all participants who received at least one dose of study drug
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
Number analyzed (Participants) | 38 | 42 | 39 | 32
Months | 6.0 [4.5 to 7.7] | 7.5 [5.6 to 11.6] | 12.0 [8.4 to NA] — NA= Not applicable as it is not evaluable. | 4.1 [3.0 to 5.9]

4. Secondary Outcome: Disease Control Rate (DCR)
Description: DCR was the percentage of the participants who had BOR of CR, PR, and stable disease (SD) with the minimum duration of SD lasting greater than or equal to 7 weeks. Only participants with measurable disease at baseline were included in evaluation of DCR, based on investigator's assessment.
Time Frame: as for outcome 2
Population: Full Analysis Set - all participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
Number analyzed (Participants) | 38 | 42 | 39 | 32
Percentage of participants | 57.9 [40.8 to 73.7] | 50.0 [34.2 to 65.8] | 48.7 [32.4 to 65.2] | 28.1 [13.7 to 46.7]

5. Secondary Outcome: Clinical Benefit Rate (CBR)
Description: CBR was the percentage of the participants who had BOR of CR, PR, and SD with the minimum duration of SD lasting greater than or equal to 23 weeks. Only participants with measurable disease at baseline were included in evaluation of CBR, based on investigator's assessment.
Time Frame: as for outcome 2
Population: Full Analysis Set - all participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
Number analyzed (Participants) | 38 | 42 | 39 | 32
Percentage of participants | 15.8 [6.0 to 31.3] | 26.2 [13.9 to 42.0] | 17.9 [7.5 to 33.5] | 6.3 [0.8 to 20.8]

6. Secondary Outcome: Number of Participants With Adverse Events (AEs)/Serious Adverse Events (SAEs) as a Measure of Safety
Description: Safety was assessed by monitoring and recording all AEs including all Common Terminology Criteria for Adverse Events (CTCAE) grades (for both increasing and decreasing severity) and SAEs; regular monitoring of hematology, clinical chemistry, and urine values; results of physical examinations, regular measurement of vital signs, and electrocardiograms (ECGs), as detailed in the Schedule of Visits and Procedures. The relationship of AEs to treatment was based on investigator judgment. Details of AEs and SAEs are provided in the reported adverse event section.
Time Frame: For each participant, from the first patient first dose till 30 days after the last dose or the cut-off date of 19 March 2013 (ie, 2.4 years)
Population: Full Analysis Set - all participants who received at least one dose of study drug
Measure: Number; unit: Participants
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
Number analyzed (Participants) | 38 | 42 | 39 | 32
Participants
  AEs | 38 | 40 | 39 | 32
  SAEs | 9 | 20 | 12 | 15

7. Primary Outcome: Progression Free Survival (PFS) Rate at Month 6
Description: PFS at Month 6 was defined as the percentage of participants who remained alive and progression-free at Month 6, based on investigator's assessment. Progression was defined using Response Assessment in Neuro-Oncology (RANO) criteria, as a greater than 25% increase in enhancing lesions despite stable or increasing steroid dose, an increase (significant) in non-enhancing T2-weighted-Fluid-Attenuated Inversion Recovery (T2/FLAIR) lesions that are not attributable to other non-tumor causes, and any new lesions. PFS rate at Month 6 was estimated from Kaplan-Meier (K-M) product-limit estimate of PFS.
Time Frame: At Month 6 from randomization (Cohort 1) or first day of treatment (Cohorts 2 and 3)
Population: Full Analysis Set included all participants who received at least one dose of study drug
Measure: Number (95% Confidence Interval); unit: Percentage of participants
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
Number analyzed (Participants) | 38 | 42 | 39 | 32
Percentage of participants | 11.0 [3.5 to 23.4] | 21.2 [10.4 to 34.5] | 8.0 [1.6 to 21.6] | 7.6 [1.3 to 21.5]

ADVERSE EVENTS:
Time Frame: For each participant, from the first patient first dose till 30 days after the last dose or the cut-off date of 19 March 2013 (ie, 2.4 years)
Description: All participants were followed for survival until death, except where a participant withdrew consent, or the Sponsor stopped the survival follow-up during the extension phase after completion of the primary study analysis. Since death was not a protocol defined reason for non-completion, the all cause mortality data below are not reflected in the Participant Flow section.
Arm/Group | Cohort 1 - Bevacizumab | Cohort 1 - Lenvatinib | Cohort 2 - Lenvatinib | Cohort 3 - Lenvatinib
All-Cause Mortality (participants affected / at risk) | 36/38 | 38/42 | 27/39 | 30/32
Serious Adverse Events (participants affected / at risk) | 10/38 | 22/42 | 12/39 | 15/32
Other Adverse Events (participants affected / at risk) | 38/38 | 40/42 | 39/39 | 31/32
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Bevacizumab (N=38) | Cohort 1 - Lenvatinib (N=42) | Cohort 2 - Lenvatinib (N=39) | Cohort 3 - Lenvatinib (N=32)
Myocardial infarction (Cardiac disorders) | 0 | 0 | 1 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 2 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 1 | 0 | 0 | 1
Intestinal perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Large intestine perforation (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 0 | 1 | 1 | 1
Pancreatitis (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Vomiting (Gastrointestinal disorders) | 0 | 2 | 0 | 1
Asthenia (General disorders) | 0 | 1 | 1 | 0
Fatigue (General disorders) | 0 | 0 | 2 | 0
General physical health deterioration (General disorders) | 0 | 2 | 0 | 0
Pyrexia (General disorders) | 0 | 1 | 0 | 0
Cholecystitis (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Hepatitis acute (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 1
Cellulitis (Infections and infestations) | 0 | 0 | 1 | 1
Diverticulitis (Infections and infestations) | 0 | 0 | 1 | 0
Perirectal abscess (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 2 | 0 | 0 | 1
Skin infection (Infections and infestations) | 0 | 1 | 0 | 0
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wound dehiscence (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 0 | 1 | 0
Lipase increased (Investigations) | 0 | 1 | 0 | 0
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 0
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 1 | 1 | 0
Myopathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Malignant neoplasm progression (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Tumour haemorrhage (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 2 | 0 | 0
Cognitive disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Convulsion (Nervous system disorders) | 2 | 5 | 1 | 2
Depressed level of consciousness (Nervous system disorders) | 0 | 1 | 1 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhage intracranial (Nervous system disorders) | 0 | 0 | 0 | 1
Haemorrhagic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
Headache (Nervous system disorders) | 0 | 1 | 2 | 0
Hemianopia homonymous (Nervous system disorders) | 0 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Peripheral motor neuropathy (Nervous system disorders) | 1 | 0 | 0 | 1
Pyramidal tract syndrome (Nervous system disorders) | 0 | 0 | 1 | 0
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 0 | 0 | 1 | 0
Confusional state (Psychiatric disorders) | 0 | 0 | 1 | 1
Delirium (Psychiatric disorders) | 0 | 0 | 0 | 1
Depressed mood (Psychiatric disorders) | 0 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Embolism (Vascular disorders) | 0 | 0 | 0 | 1
Hypertension (Vascular disorders) | 1 | 0 | 1 | 1
Hypotension (Vascular disorders) | 0 | 0 | 0 | 1
Rectal Hemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Ischaemic stroke (Nervous system disorders) | 1 | 0 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Cohort 1 - Bevacizumab (N=38) | Cohort 1 - Lenvatinib (N=42) | Cohort 2 - Lenvatinib (N=39) | Cohort 3 - Lenvatinib (N=32)
Anaemia (Blood and lymphatic system disorders) | 2 | 2 | 0 | 2
Thrombocytopenia (Blood and lymphatic system disorders) | 1 | 1 | 2 | 6
Sinus tachycardia (Cardiac disorders) | 2 | 1 | 0 | 0
Splinter haemorrhages (Cardiac disorders) | 0 | 0 | 2 | 0
Ear discomfort (Ear and labyrinth disorders) | 2 | 0 | 1 | 0
Hypoacusis (Ear and labyrinth disorders) | 0 | 0 | 0 | 2
Hypothyroidism (Endocrine disorders) | 1 | 7 | 10 | 4
Abdominal discomfort (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Abdominal distension (Gastrointestinal disorders) | 1 | 0 | 2 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 0 | 3 | 0
Abdominal pain upper (Gastrointestinal disorders) | 3 | 4 | 1 | 3
Constipation (Gastrointestinal disorders) | 6 | 7 | 9 | 6
Diarrhoea (Gastrointestinal disorders) | 7 | 7 | 11 | 10
Dry mouth (Gastrointestinal disorders) | 0 | 1 | 2 | 0
Dyspepsia (Gastrointestinal disorders) | 3 | 4 | 1 | 3
Dysphagia (Gastrointestinal disorders) | 2 | 3 | 2 | 5
Faecal incontinence (Gastrointestinal disorders) | 3 | 1 | 0 | 1
Flatulence (Gastrointestinal disorders) | 1 | 1 | 2 | 0
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 3 | 4 | 1 | 4
Gingival bleeding (Gastrointestinal disorders) | 1 | 1 | 0 | 2
Haemorrhoids (Gastrointestinal disorders) | 0 | 0 | 1 | 2
Mouth ulceration (Gastrointestinal disorders) | 1 | 0 | 2 | 1
Nausea (Gastrointestinal disorders) | 10 | 6 | 8 | 5
Oral pain (Gastrointestinal disorders) | 1 | 2 | 3 | 0
Stomatitis (Gastrointestinal disorders) | 3 | 5 | 6 | 5
Tongue ulceration (Gastrointestinal disorders) | 0 | 0 | 2 | 1
Vomiting (Gastrointestinal disorders) | 1 | 3 | 4 | 1
Asthenia (General disorders) | 1 | 1 | 1 | 2
Fatigue (General disorders) | 21 | 25 | 25 | 14
Feeling cold (General disorders) | 0 | 0 | 0 | 2
Gait disturbance (General disorders) | 5 | 5 | 1 | 2
Irritability (General disorders) | 2 | 1 | 1 | 0
Non-cardiac chest pain (General disorders) | 0 | 3 | 0 | 0
Oedema peripheral (General disorders) | 3 | 5 | 2 | 2
Candida infection (Infections and infestations) | 1 | 1 | 1 | 2
Nasopharyngitis (Infections and infestations) | 2 | 1 | 0 | 0
Oral candidiasis (Infections and infestations) | 0 | 3 | 1 | 0
Sinusitis (Infections and infestations) | 2 | 1 | 0 | 2
Tooth infection (Infections and infestations) | 1 | 0 | 2 | 0
Upper respiratory tract infection (Infections and infestations) | 2 | 2 | 0 | 1
Urinary tract infection (Infections and infestations) | 4 | 6 | 1 | 4
Contusion (Injury, poisoning and procedural complications) | 5 | 2 | 2 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 1 | 4 | 1
Alanine aminotransferase increased (Investigations) | 0 | 2 | 5 | 2
Aspartate aminotransferase increased (Investigations) | 0 | 2 | 1 | 2
Blood pressure increased (Investigations) | 3 | 2 | 2 | 2
Lipase increased (Investigations) | 0 | 1 | 2 | 2
Platelet count decreased (Investigations) | 2 | 4 | 2 | 4
Weight decreased (Investigations) | 1 | 3 | 3 | 2
Decreased appetite (Metabolism and nutrition disorders) | 3 | 9 | 6 | 3
Dehydration (Metabolism and nutrition disorders) | 0 | 2 | 3 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 5 | 7 | 4 | 2
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 4 | 0 | 3
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 3 | 0 | 4
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 1 | 0 | 3
Hypophosphataemia (Metabolism and nutrition disorders) | 1 | 1 | 2 | 3
Arthralgia (Musculoskeletal and connective tissue disorders) | 4 | 5 | 5 | 5
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 8 | 2 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 1
Muscular weakness (Musculoskeletal and connective tissue disorders) | 4 | 8 | 10 | 4
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 4 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 7 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 5 | 4 | 3 | 1
Aphasia (Nervous system disorders) | 9 | 4 | 2 | 5
Ataxia (Nervous system disorders) | 6 | 3 | 0 | 4
Balance disorder (Nervous system disorders) | 0 | 0 | 3 | 2
Cognitive disorder (Nervous system disorders) | 0 | 0 | 1 | 3
Convulsion (Nervous system disorders) | 2 | 3 | 2 | 4
Disturbance in attention (Nervous system disorders) | 0 | 3 | 0 | 0
Dizziness (Nervous system disorders) | 3 | 7 | 3 | 2
Dysarthria (Nervous system disorders) | 1 | 0 | 1 | 2
Dysgeusia (Nervous system disorders) | 0 | 3 | 1 | 1
Headache (Nervous system disorders) | 13 | 6 | 12 | 13
Hemianopia homonymous (Nervous system disorders) | 2 | 1 | 0 | 0
Hemiparesis (Nervous system disorders) | 4 | 4 | 3 | 3
Hypoaesthesia (Nervous system disorders) | 6 | 1 | 3 | 2
Memory impairment (Nervous system disorders) | 5 | 2 | 4 | 1
Paraesthesia (Nervous system disorders) | 4 | 4 | 2 | 4
Partial seizures (Nervous system disorders) | 0 | 0 | 0 | 2
Peripheral motor neuropathy (Nervous system disorders) | 3 | 0 | 0 | 2
Pyramidal tract syndrome (Nervous system disorders) | 3 | 1 | 0 | 0
Tremor (Nervous system disorders) | 0 | 1 | 4 | 1
Agitation (Psychiatric disorders) | 6 | 3 | 0 | 2
Anxiety (Psychiatric disorders) | 2 | 2 | 4 | 3
Confusional state (Psychiatric disorders) | 7 | 3 | 5 | 6
Depression (Psychiatric disorders) | 6 | 2 | 3 | 4
Flat affect (Psychiatric disorders) | 2 | 0 | 0 | 0
Insomnia (Psychiatric disorders) | 2 | 5 | 8 | 2
Mood swings (Psychiatric disorders) | 0 | 0 | 0 | 2
Glycosuria (Renal and urinary disorders) | 2 | 0 | 1 | 0
Pollakiuria (Renal and urinary disorders) | 2 | 1 | 2 | 1
Proteinuria (Renal and urinary disorders) | 2 | 6 | 4 | 9
Urinary incontinence (Renal and urinary disorders) | 3 | 4 | 4 | 2
Cough (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2 | 1
Dysphonia (Respiratory, thoracic and mediastinal disorders) | 4 | 14 | 11 | 9
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 7 | 0 | 2
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 3 | 4 | 1 | 4
Hiccups (Respiratory, thoracic and mediastinal disorders) | 2 | 2 | 3 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 0 | 0
Painful respiration (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 2
Acne (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 2 | 1 | 1 | 1
Dermatitis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Dry skin (Skin and subcutaneous tissue disorders) | 0 | 1 | 2 | 0
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 | 3 | 0 | 0
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 4 | 2 | 2 | 3
Hyperkeratosis (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 0
Night sweats (Skin and subcutaneous tissue disorders) | 1 | 0 | 2 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 1 | 3 | 3
Rash (Skin and subcutaneous tissue disorders) | 4 | 3 | 4 | 2
Deep vein thrombosis (Vascular disorders) | 2 | 0 | 1 | 0
Hypertension (Vascular disorders) | 14 | 21 | 17 | 15

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other